CLINICAL TRIAL: NCT01234545
Title: A Prospective Observational Study on the Home Treatment of Haemarthrosis With rFVIIa (Activated Recombinant Factor VII) in Haemophilia A and B Patients With Inhibitors
Brief Title: Observational Study Describing the Usual Clinical Practice Use of NovoSeven® in the Home Treatment of Joint Bleeds in Patients With Haemophilia A or B and Inhibitors
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: F7HAEM-3850; U1111-1116-2488 (Other: WHO)
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Haemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: activated recombinant human factor VII

INTERVENTIONS:
Drug: activated recombinant human factor VII — Prescription is done at the discretion of the prescribing physician as part of normal clinical routine

SUMMARY:
This trial is conducted in Africa and Asia. The aim of this study is to evaluate the efficacy of home treatment of joint bleeds (haemarthrosis) with NovoSeven® (activated recombinant human factor VII) in patients with haemophilia A and B patients with inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with congenital haemophilia and inhibitors to factor VIII or IX
* Indication of activated recombinant human factor VII for the treatment of joint bleeding located in elbow, shoulder, wrist, hip, knee, ankle

Exclusion Criteria:

* Known or suspected allergy to study product(s) or related products
* Clinically relevant coagulation disorders other than congenital haemophilia A or B

Min Age: 2 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with congenital haemophilia and inhibitors to Factor VIII or IX.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Number of bleeds managed at home | Month 8
Number of treatments resulting in the control of bleeding episode | within 9 hours after the first injection of study product
Number of treatments resulting in effective pain relief | within 9 hours after the first injection of study product

SECONDARY OUTCOMES:
Proportion of patient/caregivers with no need of any intervention from the physician to treat the bleeding episode at home | Month 8
Proportion of patients who used their entire treatment at home | Month 8

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (5):
- Algiers, Algeria
- Casablanca, Morocco
- Muscat, Oman
- Riyadh, Saudi Arabia
- Dubai, United Arab Emirates

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com